CLINICAL TRIAL: NCT02663960
Title: Is Regional Citrate Anticoagulation With Fixed Citrate Blood Concentration More Effective and Easy-to-handle Than Adjusted-dose Protocol in Adult Critically Ill Patients? A Cohort Study
Brief Title: Compare Efficacy and Simplicity of Regional Citrate Anticoagulation With Fixed Dose Versus Adjusted Citrate Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS-950
Record Dates: First submitted 2016-01-03; First posted 2016-01-26 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2016-08

CONDITIONS: Critical Illness; Kidney Replacement Disorder; Coagulation; Intravascular
Keywords: Regional citrate anticoagulation; Protocol; Filter lifespan
MeSH Terms: conditions — Critical Illness; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fixed citrate doses protocol (Experimental): Fixed citrate doses protocol: Anticoagulant Citrate Dextrose Solution ( Na+ 224, citrate 113, bicarbonate 203mmol/l, Fresenius Kabi, Italy) was administered in the prefilter ahead of the blood pump, which was set to meet a circuit citrate concentration of 4 mmol/l (duration: the maximum time is 72 hrs).
  Interventions: Other: fixed citrate doses protocol
- adjusted citrate doses protocol (Active Comparator): Adjusted citrate doses protocol: Anticoagulant Citrate Dextrose Solution ( Na+ 224, citrate 113, bicarbonate 203mmol/l, Fresenius Kabi, Italy) was administered in the prefilter ahead of the blood pump, which the starting infusion rate be set 2.5 % of blood flow ( dosage range: 160-250ml/h) and then be adjusted to obtain postfilter ionized calcium levels of less than 0.40 mmol/l (duration: the maximum time is 72 hrs. )
  Interventions: Other: adjusted citrate doses protocol

INTERVENTIONS:
Other: fixed citrate doses protocol — fixed doses of anticoagulant citrate dextrose solution to meet a circuit citrate concentration of 4 mmol/l.
  Other Names: fixed citrate circuit concentration protocol
  Arms: fixed citrate doses protocol
Other: adjusted citrate doses protocol — the starting infusion rate of anticoagulant citrate dextrose solution be set 2.5 % of blood flow and then be adjusted to obtain postfilter ionized calcium levels of less than 0.40 mmol/l.
  Arms: adjusted citrate doses protocol

SUMMARY:
Anticoagulation is required to prevent clotting in the extracorporeal circuit during continuous renal replacement therapy (CRRT). Regional citrate anticoagulation has many advantages regarding bleeding risk and filter survival. However, in clinical practice, its use worldwide has been limited by cumbersome protocols . In order to establish a simple scheme for universal application. In Aug 2015, the investigators have adopted a new protocol using a fixed citrate concentration in the filter of about 4 mmol/L (called fixed group for short) instead of conventional adjusted citrate doses according to postfilter ionized calcium levels of less than 0.4mmol/l (adjusted group), and speculated the abilities on efficacy and safety as well as convenience.

DETAILED DESCRIPTION:
Design: This study was conducted as a single-centre, cohort study. All patients older than 18 years of age who required veno-venous hemofiltration (CVVH) were consecutively screened forward (prospective) or backward (retrospective) from August, 2015 and until the expected sample size was reached.

Study protocol: Before and after implementation of a new protocol, apart from the flow rate of any supplementation (Anticoagulant-citrate-dextrose solution, 5% sodium bicarbonate injection and 10% calcium gluconate injection), CVVH was performed using same standards, including devices (Aquarius or Diapact® CRRT), venous catheter (a double lumen 12-F catheter, Arrow International Inc., USA), haemofilter (DIACAP Acute L, 2.0 m2, B. Braun Melsungen AG, Germany), commercial replacement fluids (Na+113, Cl-118, Mg++0.797, Ca++1.60, glucose 10.6mmo/l and zero bicarbonate; Qing-shan-li-kang pharmaceutical Co.,Ltd. Cheng-du, China) and Anticoagulant-citrate-dextrose solution-A (ACD-A) (Na+ 224, citrate 113, bicarbonate 203mmol/l, Fresenius Kabi, Italy) as well as monitoring algorithm. The first sample of postfilter and systemic ionized calcium was done two hours after initiation of CVVH and every six to eight hours during the first 24 hours. Afterwards, these measurements were done according to clinical needs for maintaining normal ionized calcium levels and blood pH value.

The group of fixed citrate concentration: ACD-A was administered in the prefilter ahead of the blood pump and the infusion rate was fixed and set to meet a circuit citrate concentration of 4 mmol/l. Calcium Gluconate 10% Injection was infused through the return line of the circuit and the substitution flow was initiated with 0.8 mmol calcium per liter total effluent flow and then be adjusted to obtain systemic ionized calcium levels between 0.90 and 1.2 mmol/l. Sodium bicarbonate 5% injection was infused through the return line of the circuit and the substitution flow was initiated with 3.3% of replacement fluid flow and then be adjusted to obtain blood pH value in the normal range (7.35 to 7.45)

The group of adjusted citrate doses:ACD-A was administered in the prefilter ahead of the blood pump and the starting infusion rate was 2.5 % of blood flow and then be adjusted to obtain postfilter ionized calcium levels of less than 0.40 mmol/l. Calcium Gluconate 10% Injection was infused through the return line of the circuit and the substitution flow was initiated with 7.3% of ACD-A flow, and then be adjusted to obtain systemic ionized calcium levels between 0.90 and 1.2 mmol/l. Sodium bicarbonate 5% injection was infused through the return line of the circuit and the starting infusion rate was 4% of replacement fluid flow,and then be adjusted to obtain blood pH value in the normal range (7.35 to 7.45)

Statistical analyses: groups were compared by using Fisher's exact test, Student's t test or Mann-Whitney rank-sum test as appropriate. Circuit lifetime was evaluated with Kaplan-Meier survival analysis and survival curves distribution was compared with the Log Rank test. Univariate and multivariate analysis were used to identify factors associated with mean filter lifetime in all group patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years of age who required CVVH were consecutively screened

Exclusion Criteria:

* Requiring extracorporeal membrane oxygenation (ECMO) at the time of hemofiltration, insufficient data available or missing and running time less than 6 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
the survival time of the first filter due to unexpected disconnection | the time period on CVVH, maximum 72 hour
  The interval (hours) of the installation and replacement of the first filter. The unexpected disconnection defined as filter clotting more than two grades or transmembranous pressure across the circuit exceeded >300 mmHg. The filters were changed routinely after 72 hours of CVVH treatment, so maximum survival time of the filter was recorded as 72 hrs.

SECONDARY OUTCOMES:
the overall survival time of the first filter | the time period on CVVH, maximum 72 hour
  The interval (hours) of the installation and replacement of the first filter. The survival time derived from analysis of CVVH stopping for any cause. The reasons for CVVH stopping included unexpected disconnection (defined as filter clotting more than two grades or transmembranous pressure across the circuit exceeded >300 mmHg) and expected disconnection (such as scheduled, catheter malfunction, death or discharge, metabolic complications).The filters were changed routinely after 72 hours of CVVH treatment, so maximum survival time of the filter was recorded as 72 hrs.
the frequency of change in the infusion pump rate of calcium gluconate 10% Injection | the time period on CVVH, maximum 72 hour
  recorded the change frequency (times per patient per hour ) in calcium gluconate infusion pump during the treatment period. Data were collected from records of the daily prescriptions.
the frequency of change in the infusion pump rate of Sodium Bicarbonate 5% Injection | the time period on CVVH, maximum 72 hour
  recorded the change frequency (times per patient per hour) in bicarbonate infusion pump during the treatment period. Data were collected from records of the daily prescriptions.
the frequency of change in the infusion pump rate of Anticoagulant Citrate Dextrose Solution | the time period on CVVH, maximum 72 hour
  recorded the change frequency (times per patient per hour ) in citrate infusion pump during the treatment period. Data were collected from records of the daily prescriptions.
incidences of severe metabolic disorders | the time period on CVVH, maximum 72 hour
  defined as metabolic alkalosis with blood's pH value >7.5, metabolic acidosis with blood's pH value < 7.25, hypocalcemia with ionized calcium < 0.7 mmol/L, hypercalcemia with total serum calcium ≥ 2.75mmol/L, hypernatremia with Na+ ≥ 150mmol/L), bleeding disorders (defined as the decline of hemoglobin 10g/l within 12 hours) and suspected citrate accumulation was identified as a total calcium/ionic calcium index ≥ 2.5

CONTACTS AND LOCATIONS:
Overall Officials: Bin Du, Prof., Principal Investigator — Department of medical ICU,Peking Union Medical College Hospital
Locations (1):
- MICU of Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shi Y, Qin HY, Peng JM, Hu XY, Du B. Feasibility and efficacy of modified fixed citrate concentration protocol using only commercial preparations in critically ill patients: a prospective cohort study with a historical control group. BMC Anesthesiol. 2021 Mar 30;21(1):96. doi: 10.1186/s12871-021-01319-4. PMID 33784963